CLINICAL TRIAL: NCT03146520
Title: Clinical Study for the Validation of Real Time qPCR for SDC2 Methylation in Stool DNA for Early Detection of Colorectal Cancer
Brief Title: Clinical Validation of Stool DNA-based SDC2 Methylation Test for Colorectal Cancer Detection
Status: Completed | Type: Observational
Sponsor: Genomictree, Inc. (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2016-0068
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer; Polyps; Other Cancers; Healthy
Keywords: Syndecan 2; Methylation biomarker; Colorectal cancer; EarlyTect Colon Cancer test
MeSH Terms: conditions — Colorectal Neoplasms; Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Colorectal (CRC): stage I-IV CRC subjects
  Interventions: Device: EarlyTect Colon Cancer
- Polyps: subjects with adenoma or polyps
  Interventions: Device: EarlyTect Colon Cancer
- Other cancers: subjects with other cancers
  Interventions: Device: EarlyTect Colon Cancer
- Healthy: subjects with no evidence of CRC
  Interventions: Device: EarlyTect Colon Cancer

INTERVENTIONS:
Device: EarlyTect Colon Cancer — SDC2 methylation assay by qPCR using EarlyTect Colon Cancer kit

SUMMARY:
Pivotal trials of SDC2 methylation biomarker test in stool DNA to estimate clinical sensitivity and specificity in detection of colorectal cancer.

DETAILED DESCRIPTION:
The purpose of this study is to validate the clinical performance of EarlyTect Colon Cancer test which is measuring Syndecan 2 methylation status in stool DNA to detect CRC. Syndecan 2 (SDC2) is a newly developed methylation biomarker for colorectal cancer diagnosis. Methylation status of SDC2 gene in stool DNA is determined by methylation specific qPCR. Sensitivity and specificity will be determined by comparing Stool DNA test from healthy subjects, CRC patients, and other group including polyps and other diseases.

ELIGIBILITY:
Inclusion criteria:

* sample information is complete, including sample number, gender, family history, stage of cancer, treatment history, and other disease information
* the CRC patient who has not any treatment (surgery, chemotherapy, or radiation)
* non-CRC patient who has not received any treatment (surgery, chemotherapy, or radiation) within the last 6 months
* all of above conditions are satisfied, and any one of below can be applicable; 1) confirm to be CRC with colonoscopy and/or pathological examination, 2) confirm to be inflammatory or ulcerative bowel diseases or benign hyperplastic polyp, 3) confirm to be gastrointestinal or liver cancers who are not CRC, 4) schedule to receive colonoscopy and additional confirmation test for CRC with agreement to provide the test results.

Exclusion criteria: any one of below can be applicable;

* the patient information is not complete and/or does not satisfy inclusion criteria
* the sample information is not complete and/or does not satisfy inclusion criteria
* the CRC patient who has history of colorectal cancer surgery, chemotherapy, or any other treatment
* non-CRC patient who received any chemotherapy within the last 6 months
* the patient who has limited ability or are vulnerable to accept clinical trial agreement
* the patient who is judged as not suitable for clinical trial including a psychiatric disorder by a physician

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have colorectal cancer or pre-malignancy or benign polyp or other solid tumor, or healthy normal subjects, and confirmed by colonoscopy or pathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical performance of EarlyTect Colon Cancer to detect colorectal cancer | 1.5 years
  Sensitivity and specificity of EarlyTect Colon Cancer to detect colorectal cancer (sensitivity: the ratio of positive cases in all CRC cases, specificity: the ratio of negative cases in all healthy controls)

SECONDARY OUTCOMES:
Positive ratio of SDC2 methylation in polyps | 1.5 years
  the ratio of SDC2 methylation positive in polyps
Positive ratio of SDC2 methylation in other cancers | 1.5 years
  the ratio of SDC2 methylation positive in other cancers

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh T, Kim N, Moon Y, Kim MS, Hoehn BD, Park CH, Kim TS, Kim NK, Chung HC, An S. Genome-wide identification and validation of a novel methylation biomarker, SDC2, for blood-based detection of colorectal cancer. J Mol Diagn. 2013 Jul;15(4):498-507. doi: 10.1016/j.jmoldx.2013.03.004. Epub 2013 Jun 7. PMID 23747112
- [Derived] Han YD, Oh TJ, Chung TH, Jang HW, Kim YN, An S, Kim NK. Early detection of colorectal cancer based on presence of methylated syndecan-2 (SDC2) in stool DNA. Clin Epigenetics. 2019 Mar 15;11(1):51. doi: 10.1186/s13148-019-0642-0. PMID 30876480